CLINICAL TRIAL: NCT00655720
Title: The Effects on Growth and Tolerance of Hydrolyzed Formulas Fed to Term Infants
Brief Title: The Effects on Growth of a Non-Routine Infant Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Responsible Party: Kim Merkel, Mead Johnson
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 3369-5; 3369-5
Record Dates: First submitted 2008-03-28; First posted 2008-04-10 (Estimated); Last update posted 2008-04-15 (Estimated); Status verified 2008-04

CONDITIONS: Growth
Keywords: infant formula
MeSH Terms: interventions — Infant Formula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator)
  Interventions: Other: infant formula
- 2 (Experimental)
  Interventions: Other: infant formula
- 3 (Experimental)
  Interventions: Other: infant formula

INTERVENTIONS:
Other: infant formula — 1. hydrolyzed infant formula without probiotics
  2. hydrolyzed infant formula with probiotics
  3. hydrolyzed infant formula with probiotics
  Other Names: no other names for any of the intervention arms

SUMMARY:
A study to evaluate the growth and development of term infants fed either an extensively hydrolyzed formula with probiotics, a partially hydrolyzed formula with probiotics, or an extensively hydrolyzed formula without probiotics

ELIGIBILITY:
Inclusion Criteria:

* Term infant
* Solely formula fed
* 14 days of age

Exclusion Criteria:

* History of underlying disease
* Evidence of formula intolerance
* Current illness

Ages: 12 Days to 16 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 293 (Actual)
Dates: Start 2006-03; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Growth (weight) | 106 days

SECONDARY OUTCOMES:
Tolerance | 106 days

CONTACTS AND LOCATIONS:
Overall Officials: Deolinda Scalabrin, MD, Study Director — Mead Johnson Nutrition

REFERENCES:
- [Derived] Scalabrin DM, Johnston WH, Hoffman DR, P'Pool VL, Harris CL, Mitmesser SH. Growth and tolerance of healthy term infants receiving hydrolyzed infant formulas supplemented with Lactobacillus rhamnosus GG: randomized, double-blind, controlled trial. Clin Pediatr (Phila). 2009 Sep;48(7):734-44. doi: 10.1177/0009922809332682. Epub 2009 Mar 4. PMID 19264721